CLINICAL TRIAL: NCT06070740
Title: First- Line Treatment With Durvalumab Plus XELOX Chemotherapy in Patients With Advanced Gastrointestinal Neuroendocrine Carcinoma: A Prospective Single-arm Phase II Study
Brief Title: First- Line Treatment With Durvalumab Plus XELOX Chemotherapy in Advanced Gastrointestinal Neuroendocrine Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, YueJuan Cheng, Principal investigator, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K3631
Record Dates: First submitted 2023-08-26; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Gastrointestinal Neuroendocrine Carcinoma
MeSH Terms: interventions — durvalumab; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination therapy as first-line treatment (Experimental): Durvalumab combined with XELOX chemotherapy as the first-line treatment
  Interventions: Drug: Durvalumab and Chemotherapy(oxaliplatin and capecitabine)

INTERVENTIONS:
Drug: Durvalumab and Chemotherapy(oxaliplatin and capecitabine) — Combination therapy includes:
  Durvalumab: intravenous infusion with a fixed dose of 1500 mg on day 1, repeated every 3 weeks ± 3 days; Chemotherapy: Oxaliplatin 130mg/m2 intravenous infusion on day 1, capecitabine 1000mg/m2, orally, twice a day, from day 1 to day 14; repeated every 3 weeks ± 3 days;
  After 6 cycles of combination therapy, maintain with durvalumab 1500 mg every 4 weeks ± 3 days for 2 years. Terminate the trial if confirmed disease progression, initiation of other anti-tumor therapy, unacceptable toxicity, withdrawal of informed consent or other reasons considered by the investigators.

SUMMARY:
First-Line Treatment With Durvalumab Plus XELOX Chemotherapy in Advanced Gastrointestinal Neuroendocrine Carcinoma - a prospective Single-arm Phase II Study [NCT ID not yet assigned]

DETAILED DESCRIPTION:
A prospective Single-arm Phase II Study to evaluate the effectiveness and safety of the combination treatment of durvalumab with XELOX chemotherapy as the first-line in advanced gastrointestinal neuroendocrine carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytopathologically confirmed as gastrointestinal NEC, or MiNEN (the neuroendocrine part is NEC).
* Have not previously received systemic treatment for the unresectable locally advanced or metastatic gastrointestinal NEC. Note: For patients who have previously received neoadjuvant/adjuvant or radical chemotherapy/chemoradiotherapy, the time from the end of the previous treatment to the first diagnosis of disease progression/relapse should not be less than 6 months.
* Patients with ECOG physical status score 0-1;
* The following baseline requirments must be met within 7 days before enrollment:

  1. blood tests i. Neutrophil count ≥1.5×10^9/L. ii. Hemoglobin count (HGB) ≥ 90 g/L. iii. Platelet count (PLT) ≥ 80×10^9/L.
  2. Liver and kidney function) i. Creatinine clearance ≥30ml/min.ii. Total bilirubin ≤ 1.5 ULN (Patients with biliary obstruction are allowed to be enrolled if received biliary drainage or stent implantation, and total bilirubin ≤ 2.5 × ULN).iii. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5xULN, for patients with liver metastases: ≤ 5xULN iv. Serum albumin ≥ 2.7 g/dL
* Able to provide written informed consent, and able to understand and agree to abide by the research requirements and evaluation;
* Measurable lesions according to RECIST 1.1 criteria;
* Female patients must be surgically sterilized women, postmenopausal or take high-efficiency contraception during the treatment and within 12 weeks after the treatment; male patients must be surgically sterilized men, or take high-efficiency contraception during the treatment and within 6 months after the treatment.

Exclusion Criteria:

* History of other malignant tumors in the past 5 years or at the time of enrollment (except for cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
* History of treatment with durvalumab or other PD-1/PD-L1 inhibitors; known allergies to macromolecular protein biologics, or to any ingredients of durvalumab;
* In active or history of autoimmune or inflammatory diseases (including inflammatory bowel disease, systemic lupus erythematosus, Sarcoidosis syndrome, granulomatous vasculitis, Graves disease, rheumatoid arthritis, hypophysitis, uveal inflammation, etc.);
* Received the following treatment within 2 weeks before enrollment or still in use: immunosuppressants, systemic or absorbable local hormone therapy to achieve immunosuppression (dose> 10mg/day prednisone or other equivalent steroids)
* History of abdominal fistula, gastrointestinal perforation, or abdominal abscess within 4 weeks before the start of treatment;
* History with objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, drug-related pneumonia, severe impairment of lung function, etc.;
* In active infection, including tuberculosis (evaluated by clinical assessment, including clinical history, physical examination, imaging findings, and tuberculosis examination according to the clinical practice), hepatitis B (known positive for hepatitis B virus [HBV] surface antigen [HbsAg]), Hepatitis C (HCV) or human immunodeficiency virus (human immunodeficiency virus (HIV) 1/2 antibody positive) and history of or cured HBV (defined as the presence of hepatitis B core IgG antibody and the absence of HBsAg);
* Received anti-tumor monoclonal antibody (mAb) within 4 weeks before the first use of the trialed medication, or adverse events caused by the previousl treatment have not recovered (recovery defined as ≤ grade 1 or reached the baseline level). Note: ≤2 grade neuropathy and ≤2 grade alopecia are not included. If the subject has undergone major surgery, the toxicity and/or complications caused by the surgical intervention must be fully recovered before starting treatment;
* Received live vaccines within 4 weeks before starting the treatment or may receive live vaccines during the study;
* Known history of psychotropic substance abuse, alcoholism or drug abuse;
* The subject is unable or does not agree to take the cost of self-paid examination and treatment;
* The researcher believes that it should be excluded from this study, for example, according to the researcher's evaluation, the subject has other factors that may lead to the forced termination of the study, such as other serious diseases (including mental diseases) that require combined treatment, serious abnormal laboratory results, family or social factors, which would affect the safety of the subjects or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | through study completion, an average of 1 year
  The proportion of patients who achieved complete remission or partial remission due to tumor size reduction (according to RECIST 1.1 standard)

SECONDARY OUTCOMES:
Disease Control Rate | through study completion, an average of 1 year
  The proportion of patients whose tumor shrinks and achieve complete remission, partial remission or stable condition (according to RECIST 1.1 standard);
Progression-free Survival | through study completion, an average of 1 year
  from the time of enrollment to the time of progression or death from any cause;
Overall survival time | through study completion, an average of 1 year
  from the time of enrollment to the time of death;
Adverse events | through study completion, an average of 1 year
  the frequency and severity of all adverse events (Adverse Event, AE), the severity of adverse events is evaluated according to the CTC AE v5.0 standard

CONTACTS AND LOCATIONS:
Overall Officials: Yuejuan Cheng, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China